CLINICAL TRIAL: NCT00926497
Title: Use of Procalcitonin-Guided Decision Making to Shorten Antibiotic Therapy in Suspected Neonatal Early-Onset Sepsis: Prospective Randomized Intervention Trial
Brief Title: Procalcitonin-Guided Decision Making to Shorten Antibiotic Therapy in Suspected Neonatal Early-Onset Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Martin Stocker, MD, Children's Hospital Lucerne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCTStocker
Record Dates: First submitted 2009-01-16; First posted 2009-06-23 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-05

CONDITIONS: Sepsis
Keywords: antibiotic therapy; early-onset sepsis; interventions study; procalcitonin; term and near-term neonates
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procalcitonin group (Experimental): Antibiotic therapy is discontinued when two consecutive Procalcitonin values are below predefined age-adjusted cut-off values. Antibiotic therapy could be prolonged despite fulfilled Procalcitonin criteria at the discretion of the attending physician.
  Interventions: Other: Procalcitonin-guided decision making
- Standard group (No Intervention): Standard treatment for suspected neonatal early-onset sepsis based on conventional laboratory parameters

INTERVENTIONS:
Other: Procalcitonin-guided decision making — Procalcitonin-guided decision making on duration of antibiotic therapy in suspected neonatal early onset sepsis
  Arms: Procalcitonin group

SUMMARY:
Neonatal bacterial sepsis is a major cause of mortality and morbidity and early antibiotic therapy is crucial for treatment success.

Objective: To evaluate the effect of Procalcitonin-guided decision making on duration opf antibiotic therapy in suspected neonatal early-onset sepsis.

DETAILED DESCRIPTION:
This single-centre, prospective randomized intervention study was conducted in a tertiary neonatal and paediatric intensive care unit in the Children's Hospital of Lucerne, Switzerland between June 1, 2005 and December 31, 2006. All term and near term infants with suspected early-onset sepsis were randomly assigned either to standard treatment based on conventional laboratory parameters (standard group) or to Procalcitonin-guided treatment (Procalcitonin-group). Minimum duration of antibiotic therapy was (48)-72 hours in the standard group, whereas in the Procalcitonin group antibiotic therapy was discontinued when two consecutive Procalcitonin values were below predefined age-adjusted cut-off values.

ELIGIBILITY:
Inclusion Criteria:

* Term and near-term infants with a gestational age of more than 34 weeks
* Admitted to the Children's Hospital of Lucerne, Switzerland
* Suspected neonatal early-onset sepsis
* Antibiotic therapy
* Parental consent

Exclusion Criteria:

* Surgery in the first 3 days of life
* Severe congenital malformations
* Chromosomal abnormalities

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stocker, MD, Principal Investigator — Children's Hospital Lucerne, Switzerland
Locations (1):
- children's Hospital of Lucerne, Lucerne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 1, 2005 and December 31, 2006 all term and near-term infants with a gestational age more than 34 weeks with suspected early-onset sepsis admitted to the Children's Hospital of Lucerne
Groups:
- Procalcitonin-group: Antibiotic therapy is discontinued when two consecutive PCT values are below predefined age-adjusted cut-off values.Antibiotic therapy could be prolonged despite fulfilled PCT criteria at the discretion of the attending physician.
Period: Overall Study
Arm/Group | Procalcitonin-group | Standard Group
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procalcitonin-group | Standard Group | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 61 | 121
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 39 | 36 | 75
Region of Enrollment [Number; unit: participants]
  Switzerland | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Antibiotic Treatment for More Than 72 Hours
Description: Infants treated with antibiotics for more than 72 hours (efficacy of study intervention)
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Procalcitonin-group | Standard Group
Number analyzed (Participants) | 60 | 61
participants | 33 | 55
Statistical Analysis 1: Comparison: Procalcitonin-group vs Standard Group; The trial was designed to obtain a power of 90% to detect a 30% difference between the two groups in the duration of antibiotic therapy with an estimated standard deviation of 50%; Test type: Superiority or Other; p = 0.002, Fisher Exact

2. Primary Outcome: Absolute Duration of Antibiotic Therapy
Description: Co-primary endpoint was the absolute duration of antibiotic therapy(quantitative version of the primary endpoint for estimation of effect size)
Time Frame: 1 month
Measure: Mean (Full Range); unit: hours
Arm/Group | Procalcitonin-group | Standard Group
Number analyzed (Participants) | 60 | 61
hours | 79.1 [24 to 190] | 101.5 [38 to 196]
Statistical Analysis 1: Comparison: Procalcitonin-group vs Standard Group; Test type: Superiority or Other; p = 0.012, t-test, 2 sided
Statistical Analysis 2: Comparison: Procalcitonin-group vs Standard Group; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Procalcitonin-group | Standard Group
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Procalcitonin-group | Standard Group
Secondary antibiotic therapy (Respiratory, thoracic and mediastinal disorders) | 1/60 (1) | 0/61 (0)

LIMITATIONS AND CAVEATS:
The samll sample size does not allow to prove the safety of our Procalcitonin-guided strategy. Second, because of our single center setting, our results cannot be easily be extrapolated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes